# Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

Contact Lenses with New UV-blocker Manufactured with Different Techniques

Protocol CR-6140

Version: 2.0, amendment 1

Date: 07 February 2018

Investigational Products: senofilcon A with new UV-blocker

Key Words: senofilcon A, daily wear, dispensing, subjective responses.

## Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155<sup>1</sup>, the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP)<sup>2</sup>, the Declaration of Helsinki<sup>3</sup>, and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

## **TABLE OF CONTENTS**

| | COL TITLE, NUMBER, VERSION | |
|---|---|---|
| SPONS | OR NAME AND ADDRESS | 6 |
| MEDIC | AL MONITOR | 6 |
| AUTHO | ORIZED SIGNATURES | 7 |
| CHANG | GE HISTORY | 8 |
| SYNOR | PSIS | 8 |
| COMM | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 1. IN | TRODUCTION AND BACKGROUND | 15 |
| 1.1. | Name and Descriptions of Investigational Products | 15 |
| 1.2. | Intended Use of Investigational Products | |
| 1.3. | Summary of Findings from Nonclinical Studies | 15 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5.<br>Clini | Relevant Literature References and Prior Clinical Data Relevant to cal Study | - |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 17 |
| 2.1. | Objectives | 17 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 19 |
| 3. TA | RGETED STUDY POPULATION | 20 |
| 3.1. | General Characteristics | 20 |
| 3.2. | Inclusion Criteria | 20 |
| 3.3. | Exclusion Criteria | 20 |
| 3.4. | Enrollment Strategy | 21 |
| 4. ST | UDY DESIGN AND RATIONALE | 21 |
| 4.1. | Description of Study Design | 21 |
| 4.2. | Study Design Rationale | 22 |
| 4.3. | Enrollment Target and Study Duration | 22 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | 22 |
| 5.1. | Test Article Allocation | 22 |
| 5.2. | Masking | 23 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 23 |
| 6. ST | UDY INTERVENTION | 24 |
| 6.1. | Identity of Test Articles | 24 |
| 6.2. | Ancillary Supplies/Products | 25 |

| | 6.3. | Administration of Test Articles | 25 |
|---|---|---|---|
| | 6.4. | Packaging and Labeling | 25 |
| | 6.5. | Storage Conditions | 26 |
| | 6.6. | Collection and Storage of Samples | 26 |
| | 6.7. | Accountability of Test Articles | 26 |
| 7. | STU | UDY EVALUATIONS | 27 |
| | 7.1. | Time and Event Schedule | 27 |
| | 7.2. | Detailed Study Procedures | 28 |
| | VIS | SIT 1 | 28 |
| | VIS | SIT 2 | 32 |
| | VIS | SIT 3 | 36 |
| | VIS | SIT 4 | 40 |
| | FIN | VAL EVALUATION | 42 |
| | 7.3. | Unscheduled Visits | |
| | 7.4. | Laboratory Procedures | 44 |
| 8. | SU | BJECTS COMPLETION/WITHDRAWAL | 44 |
| | 8.1. | Completion Criteria. | 44 |
| | 8.2. | Withdrawal/Discontinuation from the Study | 44 |
| 9. | PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 45 |
| 10 | ). D | EVIATIONS FROM THE PROTOCOL | 45 |
| 11 | . S' | TUDY TERMINATION | 45 |
| 12 | 2. P | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 46 |
| 13 | 3. A | DVERSE EVENTS | 47 |
| | 13.1. | Definitions and Classifications | 47 |
| | 13.2. | Assessing Adverse Events | 49 |
| | 13. | 2.1. Causality Assessment | 49 |
| | 13. | 2.2. Severity Assessment | 50 |
| | 13.3. | Documentation and Follow-Up of Adverse Events | 50 |
| | 13.4. | Reporting Adverse Events | 51 |
| | 13.4 | 4.1. Reporting Adverse Events to Sponsor | 52 |
| | | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and thorities | |
| | 13.4 | 4.3. Event of Special Interest | 53 |
| | 13.5. | Reporting of Pregnancy | 53 |
| 14 | ł. S' | TATISTICAL METHODS | 53 |

| 14 | 1.1. | General Considerations. | 53 |
|---|---|---|---|
| 14 | 1.2. | Sample Size Justification | 53 |
| 14 | 1.3. | Analysis Populations | 55 |
| 14 | 1.4. | Level of Statistical Significance | 55 |
| 14 | 1.5. | Primary Analysis | 55 |
| 14 | 1.6. | Secondary Analysis | 56 |
| 14 | 1.7. | Other Exploratory Analyses | 56 |
| 14 | 1.8. | Interim Analysis | 56 |
| 14 | 1.9. | Procedure for Handling Missing Data and Drop-Outs | 57 |
| 14 | 1.10. | Procedure for Reporting Deviations from Statistical Plan | 57 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 57 |
| 15 | 5.1. | Electronic Case Report Form/Data Collection | 57 |
| 15 | 5.2. | Subject Record | 58 |
| 16. | DA | TA MANAGEMENT | 58 |
| 16 | 5.1. | Access to Source Data/Document | 58 |
| 16 | 5.2. | Confidentiality of Information | 58 |
| 16 | 5.3. | Data Quality Assurance | 59 |
| 17. | MC | NITORING | 59 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | 59 |
| 18 | 3.1. | Study-Specific Design Considerations | 59 |
| 18 | 3.2. | Investigator Responsibility | 60 |
| 18 | 3.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 60 |
| 18 | 3.4. | Informed Consent | 61 |
| 18 | 3.5. | Privacy of Personal Data | 61 |
| 19. | STU | JDY RECORD RETENTION | 63 |
| 20. | FIN | ANCIAL CONSIDERATIONS | 63 |
| 21. | | BLICATION | |
| 22. | RE | FERENCES | 64 |
| APP | ENDI | X A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 65 |
| | | X B: PATIENT INSTRUCTION GUIDE | |
| APP | ENDI | X C: PACKAGE INSERT (APPROVED PRODUCT) | |
| APP | ENDI | X D: | 78 |
| | | LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS | 79 |
| | | EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | 87 |

| , LENS FITTING CHARACTERISTICS | 92 |
|----------------------------------------------------|-----------|
| SUBJECT REPORTED OCULAR SYMPTOMS PROBLEMS | 99 |
| FRONT AND BACK SURFACE LENS DEPOSIT GRADING P | ROCEDURE |
| DETERMINATION OF DISTANCE SPHEROCY | LINDRICAL |
| REFRACTIONS | 107 |
| , BIOMICROSCOPY SCALE | 114 |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 120 |
| PATIENT REPORTED OUTCOMES | 125 |
| WHITE LIGHT LENS SURFACE WETTABILITY | 127 |
| APPENDIX E: JJVC IRIS COLOR SCALE | 129 |
| APPENDIX F: STARTING CONTACT LENS POWER GUIDELINE | 130 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 131 |
| TABLE OF CONTENTS | |
| Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | 27 |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Contact Lenses with New UV-blocker Manufactured with Different Techniques

Protocol Number: CR-6140 Version: 2.0, amendment 1 Date: 07 February 2018

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### **MEDICAL MONITOR**

Name: John R. Buch, O.D., M.S. Title: Principal Research Optometrist

Address: 7500 Centurion Parkway, Suite 100, Jacksonville, FL 32256

Email: jbuch@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations<sup>4</sup>, ICH guidelines<sup>2</sup>, ISO 14155<sup>1</sup>, and the Declaration of Helsinki<sup>3</sup>.

| Author | See Electronic Signature Report | |
|---------------------|------------------------------------|--------|
| | John R. Buch, O.D., M.S., F.A.A.O. | DATE |
| | Principal Research Optometrist | |
| | - | |
| Clinical Operations | | |
| Manager | See Electronic Signature Report | |
| | | DATE |
| Biostatistician | See Electronic Signature Report | - |
| | | DATE |
| 5 | | |
| Data Management | See Electronic Signature Report | D.A.TE |
| | | DATE |
| Biostatistician | See Electronic Signature Report | |
| Diostatistician | See Liectronic Signuture Report | DATE |
| | | DATE |
| Reviewer | See Electronic Signature Report | |
| | | DATE |
| Approver | See Electronic Signature Report | |
| | | DATE |
| | <u> </u> | |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | John R. Buch | New document | 23 January 2018 |
| 2.0 | John R. Buch | Updates following CRRC review: • Endpoints further described • Registration status updated | 07 February 2018 |

## **SYNOPSIS**

| Protocol Title | Contact Lenses with New UV-blocker Manufactured with Different Techniques |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Phase 2b |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the Sponsor. |
| Test Article(s) | Investigational Products: Senofilcon-based contact lens containing new UV additive - often referred to as Solace. |
| Wear and Replacement<br>Schedules | Wear Schedule: Daily wear<br>Replacement Schedule: Every two weeks |
| Objectives | The primary objective of this study is to demonstrate non-inferiority of the Test lens compared to the Control lens with respect to CLUE comfort and quality of vision in order to assess Test lens performance for eventual lock on curing methodology. |

| Study Endpoints | Primary Endpoint(s): The primary endpoints are overall quality of vision and overall comfort scores using Other observation(s): Other endpoints are being evaluated chiefly to design future studies. 1. Outdoor Performance |
|---|---|
| Study Design | This study is a randomized, 4-visit, double-masked, 2x3 bilateral crossover, dispensing trial. The study lenses will be worn as daily wear (DW) for a period of two weeks each with one of the study lenses being worn twice. Each study lens is expected to be worn at least five (5) days per week for at least six (6) hours per day worn. There will be no washout period between study lenses. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations |
| Sample Size | Approximately 90 eligible subjects will be enrolled and randomized into the study. Approximately 80 subjects are targeted to complete the study. A replacement subject may be enrolled if a subject discontinues from the study prematurely; the decision whether to enroll replacement subjects will be made by the joint agreement of the Investigator and Sponsor |

| Study Duration | Subjects will wear the Test and Control lenses for two weeks each in random order with one of the study lenses being worn twice for a total of 6 weeks per subject. The enrollment will be 2 weeks, making the entire study approximately 8 weeks in duration. |
|---|---|
| Anticipated Study<br>Population | The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis. Subjects must be age 18 and older. |
| Eligibility Criteria<br>(Inclusion Criteria) | Eligibility Criteria: Potential subjects must satisfy all of the following inclusion |
| | <ol> <li>criteria to be enrolled in the study: <ol> <li>The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Healthy adult males or females age ≥18 years of age with signed informed consent.</li> <li>Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.</li> <li>The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.</li> <li>Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week.</li> <li>The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 (inclusive) in each eye.</li> <li>Have spherocylindrical best corrected visual acuity of 20/25+3 or better in each eye.</li> </ol> </li> </ol> |

## Eligibility Criteria (Exclusion Criteria)

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other bodily diseases or infections, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
- 3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear. Habitual medications taken by successful contact lens wearers are generally considered acceptable.
- 4. Habitual toric, extended wear, or multifocal contact lens wear.
- 5. Any current use of ocular medication.
- 6. Any known hypersensitivity or allergic reaction to Optifree PureMoist.
- 7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 8. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
- 9. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 10. Any active or ongoing ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
- 11. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA slit-lamp scale.
- 12. Binocular vision abnormality or strabismus.
- 13. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear.

| Disallowed<br>Medications/Interventions | Use of any prescription or over-the-counter (OTC) medications that may affect contact lens wear from 24 hours prior to receiving the study product through the study period of ~ 6 weeks. Habitual medications taken by successful soft contact lens wearers are considered acceptable. Note that habitual medications should be taken throughout the study period. |
|---|---|
| Measurements and Procedures | Subjective assessments, physiological responses, fitting characteristics. |
| Microbiology or Other<br>Laboratory Testing | None |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product for further investigation. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Opti-Free® PureMoist®, Preservative-free rewetting drops/artificial tears |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required for Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

CTP Clinical Technical Procedure

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution
MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide

| PQC | <b>Product Quality Complaint</b> |
|-----|----------------------------------|
| PRO | Patient Reported Outcome |

OA Quality Assurance OC **Quality Control** 

SAE Serious Adverse Event/Serious Adverse Experience

Statistical Analysis Plan SAP Statistical Analysis System SAS

SD Standard Deviation

SOP Standard Operating Procedure

**UADE** Unanticipated Adverse Device Effect

Unanticipated Serious Adverse Device Effect **USADE** 

VA Visual Acuity

#### INTRODUCTION AND BACKGROUND

Curing is the process used in manufacturing of contact lenses that solidifies the monomer into a lens shape. Curing is achieved at JJVC by the use of special lights assembled in a light tunnel within the manufacturing line. Historically, the lights have varied in intensity throughout the tunnel. It is unknown what happens if the manufacturing line stalls and the lens is exposed to a static curing process. A static curing process is also a more robust process and is therefore desirable provided similar clinical performance to a variable intensity process.

The present study is designed to demonstrate non-inferiority of the Test lens (static-curing process) compared to the Control lens (step-curing process) with respect to and quality of vision.

#### 1.1. Name and Descriptions of Investigational Products

This study will evaluate two senofilcon-based contact lenses containing a new UV-blocker. Both lenses are investigational. they will serve as the Control lens while the lenses manufactured with static-curing will serve as the Test lens.

## 1.2. Intended Use of Investigational Products

The intended use of the investigative product in this study is for correcting myopia and providing visual benefits in bright lighting situations. During the study, each test article will be worn bilaterally in a daily wear modality for at least 6 hours per day and 5 days per week for approximately two weeks each. The subject will wear either the test or control article twice and the other study article once.

## 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding senofilcon A with new UV-blocker, refer to the latest version of the Investigator's Brochure.

## 1.4. Summary of Known Risks and Benefits to Human Subjects

The risks of wearing soft contact lenses are well known and are described in the Investigator's Brochure and Informed Consent. The material safety testing/lens release criteria was determined based on the Risk Assessment. Benefits to the subjects include the correction of their refractive error with the potential of improved 'visual comfort' in bright lighting environments.

For the most comprehensive risk and benefit information regarding senofilcon A with new UV-blocker, refer to the latest version of the Investigator's Brochure.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study



The literature is absent of any articles pertaining to soft contact lenses containing the new type of UV blocker. A list of relevant literature references pertaining to glare, eyestrain, and light filtering is provided:

- 1 Agarwal, S., Goel, D., & Sharma, A. (2013). Evaluation of the factors which contribute to the ocular complaints in computer users. J Clin Diagn Res,7(2), 331-335.
- 2 Eperjesi, F., Fowler, C. W., & Evans, B. J. (2002). Do tinted lenses or filters improve visual performance in low vision? A review of the literature. Ophthalmic and Physiological Optics, 22(1), 68-77.
- 3 Hickcox, K. S., Narendran, N., Bullough, J. D., & Freyssinier, J. P. (2013). Effect of different coloured luminous surrounds on LED discomfort glare perception. Lighting Research and Technology, 1477153512474450.
- 4 Leguire, L. E., & Suh, S. (1993). Effect of light filters on contrast sensitivity function in normal and retinal degeneration subjects. Ophthalmic and Physiological Optics, 13(2), 124-128.

- Morse, R. S. (1985, October). Glare filter preference: influence of subjective and objective indices of glare, sharpness, brightness, contrast and color. In Proceedings of the Human Factors and Ergonomics Society Annual Meeting (Vol. 29, No. 8, pp. 782-786). SAGE Publications.
- 6 Pérez-Carrasco, M. J., Puell, M. C., Sánchez-Ramos, C., López-Castro, A., & Langa, A. (2005). Effect of a yellow filter on contrast sensitivity and disability glare after laser in situ keratomileusis under mesopic and photopic conditions. Journal of Refractive Surgery, 21(2), 158-165.
- 7 Sheedy, J. E., Hayes, J., & ENGLE, J. (2003). Is all asthenopia the same? Optometry & Vision Science, 80(11), 732-739.
- 8 Steen, R., Whitaker, D., Elliott, D. B., & Wild, J. M. (1994). Age-related effects of glare on luminance and color contrast sensitivity. Optometry & Vision Science, 71(12), 792-796.
- 9 Vincent, A. J., Spierings, E. L., & Messinger, H. B. (1989). A controlled study of visual symptoms and eye strain factors in chronic headache. Headache: The Journal of Head and Face Pain, 29(8), 523-527.
- 10 Wilkins, A. J., & Evans, B. J. (2010). Visual stress, its treatment with spectral filters, and its relationship to visually induced motion sickness. Applied Ergonomics, 41(4), 509-515.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

## 2.1. Objectives

Primary Objective(s)

The primary objective of this study is to compare the clinical performance of two study contact lenses using different curing techniques with respect to CLUE comfort and vision.

Other Objectives(s)

Other objectives of this study are to compare the clinical performance of two study contact lenses using different curing techniques with respect to driving, indoor and outdoor performance items, CLUE handling and the rate of Grade 3 or higher slit lamp findings.

## 2.2. Endpoints

Primary Endpoint(s)

#### **CLUE Comfort and Vision**

The primary endpoints are overall quality of vision and overall comfort scores using Contact Lens User Experience (CLUE)<sup>TM</sup> questionnaire at the two-week follow-up. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.

#### Other Observation(s)

Other endpoints are being evaluated chiefly to design future studies.

## 1. <u>Driving Performance</u>

Driving performance will be assessed by two individual patient reported outcome (PRO) questions at the 2-week follow-up evaluation. The individual items are as follows:

- A. Reduction in glare while driving during the day (Item ID: MIS00617)
- B. Reduction in glare while driving during the night (Item ID: MIS00618)

#### 2. <u>Indoor Performance</u>

Indoor performance will be assessed by three individual patient reported outcome (PRO) questions at the 2-week follow-up evaluation. The individual items are as follows:

- A. Reduction in glare from the computer screen (Item ID: MIS00628)
- B. Reduction in glare caused by bright indoor lights (Item ID: MIS00625)
- C. Reduction in glare caused by bright light coming through the window (Item ID: MIS00626)

#### 3. Outdoor Performance

Outdoor performance will be assessed by four individual patient reported outcome (PRO) questions at the 2-week follow-up evaluation. The individual items are as follows:

- A. Ability to see comfortably in bright sunlight (Item ID: MIS00613)
- B. Reduction in glare in bright sunlight (Item ID: MIS00614)
- C. Reduction in squinting in bright sunlight (Item ID: MIS00615)
- D. Reduction in eye strain in bright sunlight (Item ID: MIS00616)

All driving, indoor and outdoor (PRO) items above will be assessed using the same excellence scale of; 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor.

#### 4. CLUE Handling

Handling scores will be assessed by using Contact Lens User Experience (CLUE)<sup>TM</sup> questionnaire at the two-week follow-up.

5. Physiological Response assessed at each visit.

# 2.3. Hypotheses

Primary Hypotheses

| Primary Hypotheses | |
|---|---|
| Endpoint | Hypothesis |
| Overall CLUE Vision | The test lens will be non-inferior to the control lens at the 2-week follow-up with respect to CLUE overall quality of vision. A non-inferiority margin of -5 points will be used. |
| Overall CLUE Comfort | The test lens will be non-inferior to the control lens at the 2-week follow-up with respect to CLUE overall comfort. A non-inferiority margin of -5 points will be used. |

Both Primary hypotheses must be met for this study to be considered successful.

Other Hypotheses

| | Other Hypotheses |
|---|---|
| Endpoint | Hypothesis |
| Outdoor Performance<br>Measures | The test lens will be superior to the control lens in at least 2 of the following 4 outdoor performance measure(s) at the 2-week follow-up. An odds ratio margin of 1 will be used. 1. Ability to see comfortably in bright sunlight 2. Reduction in glare in bright sunlight 3. Reduction in squinting in bright sunlight 4. Reduction in eye strain in bright sunlight |
| Driving Performance<br>Metrics | The test lens will be non-inferior to the control lens in both of the following driving performance metrics at the 2-week follow-up. An odds ratio margin of 0.67 will be used. 1. Reduction in glare while driving during the day 2. Reduction in glare while driving during the night |
| Indoor Performance<br>Measures | The test lens will be superior to the control lens in at least 2 of the following 4 outdoor performance measure(s) at the 2-week follow-up. An odds ratio margin of 1 will be used. 1. Reduction in squinting while working on the computer 2. Reduction in glare from the computer screen 3. Reduction in glare caused by bright indoor lights 4. Reduction in glare caused by bright light coming through the window |
| CLUE Handling | CLUE handling of the step-cure and static cure lenses will be no different from each other. |
| Physiological Response | Physiological responses of the step-cure and static cure lenses will be no different from each other. |

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Approximately 90 subjects will be enrolled to ensure that at least 80 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of 18 or older. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. Subjects will wear the test and control contact lenses approximately two weeks each on a daily wear (DW) basis, then wear either the test or control lens again for two weeks, for a total study duration of approximately 42 days (6 weeks) per subject.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria after Screening

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Healthy adult males or females age ≥18 years of age with signed informed consent.
- 4. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.
- 5. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.
- 6. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week.

#### Inclusion Criteria after Baseline

- 7. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 (inclusive) in each eye.
- 8. The subject's refractive cylinder must be  $\leq$  -1.00 D in each eye.
- 9. Have spherocylindrical best corrected visual acuity of 20/25+3 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other bodily

- diseases or infections, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
- 3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear. Habitual medications taken by successful contact lens wearers are generally considered acceptable.
- 4. Habitual toric, extended wear, or multifocal contact lens wear.
- 5. Any current use of ocular medication.
- 6. Any known hypersensitivity or allergic reaction to Optifree PureMoist.
- 7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
- 8. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
- 9. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).

#### Exclusion Criteria after Baseline

- 10. Any active or ongoing ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
- 11. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA slit-lamp scale.
- 12. Binocular vision abnormality or strabismus.
- 13. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

## 4.1. Description of Study Design

This study is a randomized, 4-visit, double-masked, 2x3 bilateral crossover, dispensing trial. Approximately 90 subjects will be screened and enrolled to ensure that at least 80 subjects to complete.

The study begins with an initial visit (Visit 1). If a subject is found to meet all eligibility criteria, they will be random to one of two lens wear sequences (Test/Control/Control or Control/Test/Test).

If the subject is dispensed study lenses at the initial visit, 3 follow-up visits will be conducted. The follow-up visits occur approximately 2, 4 and 6 weeks after the initial visit. Unscheduled follow-up visits may occur during the study. Subjects will be advised to wear the study lenses at least five (5) days per week for at least six (6) hours per day for a period of two weeks each. Lens replacement is scheduled at 2 and 4-week follow-up visits.

## 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. This design was considered since the study period is relatively short the design can be cost effective and more efficient comparisons between treatments can be made than compared a parallel study since fewer subjects are required to achieve the same pre-specified statistical power.

Therefore, this study utilizes a high order 3-period by 2-treatment crossover design to estimate the true effect of the Test lens without any potential bias from the carry-over effect.

## 4.3. Enrollment Target and Study Duration

Approximately 90 subjects will be enrolled to ensure that at least 80 subjects will complete the study. Enrolled subjects will be habitual wearers of spherical contact lenses. All subjects will be the age of 18 or older. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them. Subjects will wear the Test and Control contact lenses approximately two weeks each on a daily wear (DW) basis, then wear either the Test or Control lens again for two weeks, for a total study duration of approximately 42 days (6 weeks) per subject.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

Use of the test articles will be randomized using a randomization scheme supplied by the study biostatistician.

This is a multi-site, double-masked, dispensing and randomized study. The study lenses will be worn in a bilateral and random fashion using a 2 treatment by 3 period (2x3) crossover design.

A block size of two (2) sequences will be utilized. A computer-generated randomization scheme will be used to randomly assign subjects, in blocks of 2, to one of the two possible lens wear sequences (TEST/CONTROL/CONTROL or CONTROL/TEST/TEST). The random scheme will be generated by site using the PROC PLAN procedure from SAS Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment according to the randomization list and not pre-select or assign subjects. The randomized

assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected.

#### 5.2. Masking

Both test lenses will contain the same new UV-blocker. Therefore, double-masking is possible and will be used to keep both the subject and investigators masked to the identity of the study lenses throughout the duration of the study period. Every attempt will be made to keep the other clinical trial personnel involved in the study (e.g. Data management and Biostatistician) unaware of the identity of the study lenses.

The identity of the study lenses will be masked by over labeling the blister packs with a label containing the study number, lot number, sphere power, expiration date and the randomization codes P or W. Only the personnel involved in the over labeling and the unmasked statistician will have access to the lens decode information translating the randomization codes into test and control groups. The medical monitor will also have access to the decode information in case breaking the mask is necessary for the urgent medical treatment of a subject.

Masking will be used to reduce potential bias. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will be masked as to the identity of the investigational product.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued will be replaced.

## 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- Investigator or designee (documented on the Delegation Log) will consult the lens
  fitting schedule/randomization scheme to obtain the test article assignment for that
  subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 6. STUDY INTERVENTION

### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test | Control |
|---|---|---|
| Name | ECL100 | ECL100 |
| Manufacturer | JJVC | JJVC |
| Lens Material | senofilcon A | senofilcon A |
| Nominal Base Curve @ 22°C | 8.4 | 8.4 |
| Nominal Diameter @ 22°C | 14.0 | 14.0 |
| Nominal Distance Powers (D) | -1.00 to -6.00 in 0.25<br>steps | -1.00 to -6.00 in 0.25<br>steps |
| Water Content (Optional) | 38 | 38 |
| Center Thickness (Optional) | 0.085 | 0.085 |
| Oxygen Permeability (Dk) | 103 | 103 |
| Modality in Current Study | Daily wear | Daily wear |
| Replacement Frequency | 2 weeks | 2 weeks |
| Packaging Form (vial, blister, etc.) | Sterile blister pack | Sterile blister pack |
| Curing Light Source Bulb Type | LED | LED |
| Hydration | PG | PG |
| Cure Technique | Static | Step |

Approximately 25 lenses per sku will be made available based on the following factors: sample size, 2x3 design, bilateral wear, biweekly replacement, safety margin of 2x, and US distribution model for the range of lenses -1.00 through -6.00 D.

## 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Solution | |
|---|---|---|
| Solution Name /<br>Description | Opti-Free® PureMoist® | Eye-Cept Rewetting<br>Drops |
| Lot Number or Other<br>Identifier | Varies | Varies |
| Manufacturer | Alcon Laboratories, Fort Worth, TX | Optics Laboratories |
| Maximum<br>Preservative | 0.001% polyquaternium-1, 0.0006% myristamidopropyl dimethylamine | NA |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

## 6.4. Packaging and Labeling

The test articles will be packaged in blisters as the primary packaging. The test article will be over-labeled to mask the subject/Investigators to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:

## 6.5. Storage Conditions

All worn study lenses will be collected from the subject, placed in labeled glass vials with Opti-Free® Puremoist®, and stored refrigerated or frozen until they are shipped back to the Sponsor. The lenses will be shipped in special containers to keep the lenses refrigerated.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

All worn study lenses will be collected from the subject, placed in labeled glass vials with Opti-Free® Puremoist®, and stored refrigerated or frozen until they are shipped back to the Sponsor. The lenses will be shipped in special containers to keep the lenses refrigerated.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

## 6.6. Collection and Storage of Samples

All worn lenses will be collected and stored in a labeled vial. The lenses will be stored cold at the investigational site and shipped back to JJVC cold for lab testing.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

## 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

## 7. STUDY EVALUATIONS

## 7.1. Time and Event Schedule

Table 3: Time and Events

| Procedure | Baseline | Trial Fit & Dispense | Follow-up | Unsched | Exit |
|---|---|---|---|---|---|
| Visit | 1 | 1, 2, 3 | 2, 3, 4 | PRN | 4 |
| Visit Window | - | - | 13-15<br>Days | - | - |
| Informed consent | ✓ | - | - | - | - |
| Eligibility screening | ✓ | - | - | - | - |
| CLUE Baseline Questionnaire | <b>√</b> | 1 | - | - | - |
| GSI Background Questionnaire | | | | | |
| Other Questionnaires | ✓ | - | - | - | - |
| Subject demographics | ✓ | - | - | - | - |
| General health and medication history | <b>✓</b> | - | - | - | - |
| Subject's own contact lens information | <b>✓</b> | - | - | - | - |
| Habitual lens care | ✓ | - | - | - | - |
| Entrance visual acuity | ✓ | - | - | - | - |
| Spherocylindrical refraction and BVA | <b>✓</b> | - | - | <b>√</b> | ✓ |
| Slit lamp biomicroscopy | ✓ | - | ✓ | <b>√</b> | - |
| Expanded Conjunctival<br>Redness | <b>✓</b> | - | ✓ | ✓ | - |
| Expanded Corneal Staining | ✓ | - | ✓ | ✓ | - |
| Trial fitting lens information | - | ✓ | - | - | - |
| Lens Damage | - | ✓ | - | - | - |
| Distance spherical over-<br>refraction | - | ✓ | <b>√</b> | - | - |
| Lens modification | - | ✓ | - | - | - |
| Visual acuity | - | <b>√</b> | ✓ | <b>√</b> | - |
| Lens fitting assessment | - | <b>√</b> | ✓ | * | - |
| Lens wettability | - | ✓ | ✓ | * | - |
| Lens dispensing information and criteria | - | ✓ | - | - | - |

| Procedure | Baseline | Trial Fit &<br>Dispense | Follow-up | Unsched | Exit |
|---|---|---|---|---|---|
| Visit | 1 | 1, 2, 3 | 2, 3, 4 | PRN | 4 |
| Visit Window | - | - | 13-15<br>Days | - | - |
| Patient instructions | - | <b>✓</b> | - | - | - |
| Lens information | - | 1 | ✓ | ✓ | - |
| Compliance | - | - | ✓ | ✓ | - |
| Wearing times | - | - | ✓ | ✓ | - |
| CLUE Follow-Up<br>Questionnaire | - | - | ✓ | * | - |
| GSI Product Performance<br>Questionnaire | - | - | <b>✓</b> | * | - |
| Symptoms | - | ✓ | ✓ | ✓ | - |
| Lens preference | - | - | V 2, 3, 4 | - | - |
| Surface characteristics | - | - | <b>√</b> | * | - |
| Chief complaint, diagnosis, treatment | - | - | - | ✓ | - |
| * if wearing study contact lenses | | | | | |

# 7.2. Detailed Study Procedures

VISIT 1
Subjects must enter Visit 1 wearing their habitual contact lenses.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's date of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Baseline<br>Questionnaires | The subject will respond to the following questionnaires: 1. CLUE Baseline Questionnaire |
| 1.7 | Other<br>Questionnaires | The subject will respond to additional questionnaires: 1. Activity History |
| 1.8 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.9 | Remove Habitual<br>Lens | The subject's habitual lenses will be removed and stored in their own lens case. If they forgot to bring their lens case, one will be provided to them. |
| 1.10 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale ( |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. | |
| 1.11 | Iris Color | The investigator will record the subject's iris color based on the scale provided. | Appendix E |
| 1.12 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform subjective best sphere refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use a balancing technique (e.g., the duochrome test for binocular balancing, or the binocular blur balancing test, etc.,) and record the best corrected distance visual acuity (OD, OS, and OU) to the nearest letter. | |
| 1.13 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.14 | Lens Fitting | The Lens Randomization Table will be used to determine which study lens is worn second. The lens powers are based on the vertexed (12mm), spherical equivalent subjective refraction. The investigator or subject will place the lenses on. Quickly check for any lens damage and replace if necessary. |
| 1.15 | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 1.16 | Spherical Over-<br>refraction &<br>Optimization | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. |
| 1.17 | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.18 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.19 | GSI Post-Fit<br>Questionnaire | Subjects will respond to the GSI Post-Fit Questionnaire. |
| 1.20 | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 1.21 | Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement edge lift excessive movement in primary and up gaze insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up Note: if lens fit is unacceptable subject will be discontinued from the study. |
| 1.22 | Lens Wettability | Record the white light lens wettability of both lenses. |
| 1.23 | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.24 | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>A patient instruction booklet will be provided.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> <li>Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit).</li> <li>Note 2: The subject's habitual contact lenses cannot be worn at any time during the study.</li> </ol> |

## VISIT 2

The follow-up will occur 13-15 days after the initial dispensing. The subjects must enter the visit wearing their study contact lenses.

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| 2.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule and cleaning regime. Outdoor and total hours will be asked. |
| 2.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.5. | Follow-Up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance | |
| 2.6. | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | 5 |
| 2.7. | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Imbal exposure at primary gaze or with extreme eye movement edge lift excessive movement in primary and up gaze insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up Note: if lens fit is unacceptable subject will be discontinued from the study. | |
| 2.8. | Surface Deposits | Record any front and back surface lens deposits. | |
| 2.9. | Wettability<br>Characteristics | Record the white light lens wettability of both lenses. | |
| 2.10. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with OptiFree PureMoist. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV. | |

| Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| 2.11. | Slit Lamp<br>Biomicroscopy | Slit Lamp Classification Scale (CTP-2018) will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings (CTP-2002) and Corneal Staining Assessment (CTP-2003) will be emphasized using a more detailed scale. Note: Findings must be Grade 0, 1 or 2 as graded on the FDA scale (CTP-2018) to continue onto Trial Period 2. If the subject is not eligible (Grade 3 or 4), they must be followed as an adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors immediately. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

| Visit 2: Treatment 2 Lens Fitting | | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.12. | Lens Fitting | The Lens Randomization Table will be used to determine which study lens is worn second. The lens powers are based on the vertexed (12mm), spherical equivalent subjective refraction. The final lens power from Trial Fitting 1 can also be used. The investigator or subject will place the lenses on. Quickly check for any lens damage and replace if necessary. | Appendix F |
| 2.13. | Lens Settling | Please wait at least 5 minutes before continuing. | |
| 2.14. | Spherical Over-<br>refraction &<br>Optimization | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. | |
| 2.15. | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. | |
| 2.16. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |

| | Visit 2: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 2.17. | GSI Post-Fit<br>Questionnaire | Subjects will respond to the GSI Post-Fit Questionnaire. |
| 2.18. | Visual Acuity | Record the distance visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 2.19. | Lens Fit Assessment | The fit of the lens is judged by the investigator as pass or fail based on the criteria below. If the fit of the lens is judged as a failure, the subject is terminated from the study. To be judged as a failure, the lens must display one or more of the following: 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 2.20. | Lens Wettability | Record the white light lens wettability of both lenses. |
| 2.21. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |
| 2.22. | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days.</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥ 6 hours per day, ≥ 5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> </ol> |

| Visit 2: Treatment 2 Lens Fitting | | |
|---|---|---|
| Step | Procedure | Details |
| | | Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit). Note 2: The subject's habitual contact lenses cannot be worn at any time during the study. |

## VISIT 3

The follow-up will occur 13-15 days following Visit 2. The subjects must enter the visit wearing their study contact lenses.

| Visit 3: Treatment 2 Follow-Up 1 | | | |
|---|---|---|--|
| Step | Procedure | Details | |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications<br>Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. | |
| 3.2. | Wearing Time | Record the average wearing time and comfortable wearing time. | |
| 3.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. | |
| 3.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.5. | Follow-up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance | |
| 3.6. | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |
| 3.7. | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. | |
| | Visit 3: Treatment 2 Follow-Up 1 | | | |
|---|---|---|--|--|
| Step | Procedure | Details | | |
| | | An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or | | |
| | | <ul> <li>with extreme eye movement</li> <li>edge lift</li> <li>excessive movement in primary and</li> </ul> | | |
| | | <ul> <li>up gaze</li> <li>insufficient movement in all three of<br/>the following conditions: primary<br/>gaze, up gaze, and Josephson push<br/>up</li> </ul> | | |
| | | <b>Note:</b> if lens fit is unacceptable subject will be discontinued from the study. | | |
| 3.8. | Surface Deposits | Record any front and back surface lens deposits. | | |
| 3.9. | Lens Wettability | Record the white light lens wettability of both lenses. | | |
| 3.10. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVC for 45 days after LSLV for laboratory testing (Section 7.4). | | |

| | Visit 3: Treatment 2 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 3.11. | Slit Lamp Findings | Slit Lamp Classification Scale will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings and Corneal Staining Assessment will be emphasized using a more detailed scale. Note: Findings must be Grade 0, 1 or 2 as graded on the FDA scale (CTP-2018) to continue onto Trial Period 2. If the subject is not eligible (Grade 3 or 4), they must be followed as an adverse event. Once resolved, the subject is terminated from the study. Adverse events must be reported to the JJVC monitors immediately. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

| | Visit 3: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Step Procedure Details | |
| 3.12. | Lens Fitting | The Lens Randomization Table will be used to determine which study lens is worn third. The lens powers are based on the vertexed (12mm), spherical equivalent subjective refraction. The final lens power from Trial Fitting 1 or 2 can also be used. The investigator or subject will place the lenses on. Quickly check for any lens damage and replace if necessary. |
| 3.13. | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 3.14. | Spherical Over-<br>refraction &<br>Optimization | Perform a spherical over-refraction OD and OS. Optimize the lens power to achieve an over-refraction of ±0.00 D OD and OS. Ensure that any new lenses are not damaged. One modification attempt will be allowed. |
| 3.15. | Time Interval | Please wait for at least 10 minutes from final lens insertion to continue. |
| 3.16. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |

| | Visit 3: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 3.17. | GSI Post-Fit<br>Questionnaire | Subjects will respond to the GSI Post-Fit Questionnaire. |
| 3.18. | Visual Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Smaller lines must be shown until the subject incorrectly identifies at least 50% of the letters. |
| 3.19. | Lens Fit Assessment | Subjective Assessment of the Lens Fit. If the fit is graded as unacceptable based on the criteria below, then the subject is discontinued from the study and will not be replaced. 1. Limbal exposure in any gaze 2. Edge lift 3. Insufficient and/or excessive movement in all three movement categories |
| 3.20. | Lens Wettability | Record the white light lens wettability of both lenses. |
| 3.21. | Continuance | For the subject to continue in the study, they must meet all three of the following criteria: 1. Visual acuity is 20/30 or better OD and OS 2. The lens fit is acceptable OD and OS 3. Investigator approval. If the Investigator does not approve the dispensing of the first study lens, then the study is terminated for that subject. |

| | Visit 3: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 3.22. | Dispense | <ol> <li>The lenses will be dispensed for 13-15 days.</li> <li>The subjects should wear their lenses similar to the inclusion criteria: ≥6 hours per day, ≥5 days per week.</li> <li>The lenses will be worn as daily wear only.</li> <li>All subjects will be provided Opti-Free® PureMoist® to be used in a rub regime.</li> <li>Preservative-free rewetting drops are permitted if needed.</li> <li>The lenses must be stored in the supplied case out of direct sunlight.</li> <li>Note 1: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement (extra lenses cannot be given at the dispensing visit).</li> <li>Note 2: The subject's habitual contact lenses cannot be worn at any time during the study.</li> </ol> |

# VISIT 4

The follow-up will occur 13-15 days after the dispensing of the second study lenses. The subjects must enter the visit wearing their study contact lenses.

| | Visit 4: Treatment 3 Follow-Up 1 | |
|---|---|---|
| Step | Step Procedure Details | |
| 4.1. | Adverse Events and<br>Concomitant<br>Medications<br>Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 4.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 4.3. | Compliance | Confirm compliance with the prescribed wear schedule. Outdoor and total hours will be asked. |
| 4.4. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-<br>ended symptoms questionnaire. |

| | Visit 4: Treatment 3 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 4.5. | Follow-up<br>Questionnaire | Subjects will respond to the following questionnaires: 1. CLUE Follow-up 2. GSI Product Performance |
| 4.6. | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity with the contact lenses (OD, OS, and OU) to the nearest letter. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 4.7. | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: • limbal exposure at primary gaze or with extreme eye movement • edge lift • excessive movement in primary and up gaze • insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up Note: if lens fit is unacceptable subject will be discontinued from the study. |
| 4.8. | Surface Deposits | Record any front and back surface lens deposits. |
| 4.9. | Lens Wettability | Record the white light lens wettability of both lenses. |
| 4.10. | Lens Removal &<br>Storage | Both lenses will be removed and stored wet in a labeled container with Opti-Free® PureMoist®. The lenses can be stored refrigerated or frozen prior to shipment back to the Sponsor. Lenses will be stored at JJVCI for 45 days after LSLV for laboratory testing (Section 7.4). |

| Visit 4: Treatment 3 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| 4.11. | Slit Lamp Findings | Slit Lamp Classification Scale (will be used to grade the findings. Record only whole numbers. Limbal and Bulbar Conjunctival Hyperemia findings (and Corneal Staining Assessment) will be emphasized using a more detailed scale. Note: Findings must be Grade 0, 1 or 2 as graded on the FDA scale to continue onto Trial Period 2. If the subject is not eligible (Grade 3 or 4), they must be followed as an adverse event. Adverse events must be reported to the JJVC monitors immediately. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details CTP |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Subjective Perform bare-eye subjective spherocylindrical refraction with a phoropter | |

### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications

- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Step | Procedure | Details |
|---|---|---|
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Change of Medical<br>History and<br>Concomitant<br>Medications | Questions regarding the change of subjects' medical history and concomitant medications. |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |
| U.4 | Subjective Sphero-<br>cylindrical<br>Refraction | The investigator will complete a subjective refraction (sphere and cylinder) and record the resultant distance visual acuity OD, OS, and OU to the nearest letter. |
| U.5 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If no slit lamp finding is noted on the EDC form it is considered as a zero "0" Grade for all observations listed. After the slit lamp examination, at the discretion of the Investigator, rinse the |
| | | subject's eyes thoroughly with preservative-<br>free saline. |
| U.6 | Dispensing (if applicable) | Additional lenses may be dispensed if one is lost or torn during the wearing period. |
| U.7 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS and OU) to the nearest letter. |

## 7.4. Laboratory Procedures

The optical bench will be used to measure the light transmission characteristics for all worn Test lenses. The findings are for internal information only and will not be part of the final report.

### 8. SUBJECTS COMPLETION/WITHDRAWAL

### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- completed all scheduled visits

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol (e.g. Subject more than 2 days out of visit window).
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear (subjects missing more than 2 days of missed lens wear within a period 1 of week should be discontinued)
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed any scheduled study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject will be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to

follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: see Section 3.3.

Concomitant therapies that are disallowed include: see Section 3.3.

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this

protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

**Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity (BSCVA) equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions

• Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation <2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

**Unanticipated Adverse Device Effect (UADE)** – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 0)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g.

- concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset

- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

### 13.4.1. Reporting Adverse Events to Sponsor

# Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

### 13.4.3. Event of Special Interest

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

# 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4, add/modify software if necessary (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

### 14.2. Sample Size Justification

This study was designed and powered to show non-inferiority between the Test lens compared to the Control lens with respect to CLUE comfort and vision. It was assumed there was no difference between the Test and Control lenses. The sample size was calculated to achieve a minimum statistical power of 90% and a type I error of 5%.

The sample size calculation was based on historical data from a similar study, CR-5960 The Test lens from CR-5960 is the Control for this study. CR-5960 enrolled 133 subjects, of which 130 (97.7%) were dispensed study lenses. Of the dispensed subjects, 127 (95.5%) completed the study and 3 (2.3%) subjects were discontinued. The per-protocol population included 121 (91.0%) subjects out of the total 127 that completed. Table 4 summarizes CLUE scores from CR-5960 at the 2-week follow-up.<sup>13</sup>

Table 4: Descriptive CLUE scores from CR-5960 (Historical Data)

| CLUE Domain | Study Lenses | |
|---|---|---|
| | Acuvue Oasys | Solace – 25% differential |
| Comfort [mean (SD <sup>1</sup> )] | 61.185 (24.2024) | 64.339 (24.2132) |
| Vision [mean (SD <sup>1</sup> )] | 66.792 (20.0073) | 69.445 (20.1752) |

<sup>&</sup>lt;sup>1</sup>SD: Standard Deviation

Sample size calculation for CLUE comfort and vision were carried out using an approximation of the power of an F-test derived from the non-centrality parameter calculated form the observed F-statistic of a linear model. <sup>14</sup>

### Model details:

CLUE comfort and vision were analyzed separately using a linear mixed model. Lens type, was included as the only fixed effect. A compound symmetric (CS) covariance was used to model the correlation between measurements within the same subject across study periods. Below is the variance-covariance matrix used in the CLUE each model.

$$\sum_{comfort} \begin{pmatrix} 349.3 & 110.9 & 110.9 \\ 110.9 & 349.3 & 110.9 \\ 110.9 & 110.9 & 349.3 \end{pmatrix}$$

$$\sum_{vision} \begin{pmatrix} 257.4 & 82.1 & 82.1 \\ 82.1 & 257.4 & 82.1 \\ 82.1 & 82.1 & 257.4 \end{pmatrix}$$

**Table 5: Sample Size Calculations for CLUE Comfort and Vision** 

| <b>CLUE Domain</b> | Number to Complete | Power (%) |
|--------------------|--------------------|-----------|
| Comfort | 50 | 77% |
| | 60 | 85% |
| | 80 | 93% |
| Vision | 50 | 88% |
| | 60 | 93% |
| | 80 | 98% |

Assuming no difference between the Test lens and Control lens, the sample size required to achieve non-inferiority with a minimum power of 90% and a type I error controlled at 5% was estimated to be 80 subjects.

# 14.3. Analysis Populations

### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

# **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

# 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

# 14.5. Primary Analysis

### **CLUE** Comfort and Vision

Overall comfort and vision CLUE scores will be analyzed separately using a linear mixed model adjusting for baseline values as a covariate. Sequence of lens wear, period, lens type, first order carryover effect will be included in each model as fixed effects. An appropriate covariance structure will be used to model the residual errors between measurements within same subject across study periods (R-side). The covariance structure will be selected based on the finite-sample corrected Akaike's Information Criterion. Covariance structures considered include:

- Unstructured Covariance Structure (UN)
- Homogenous Compound symmetry (CS)
- Heterogeneous Compound Symmetry (CSH)
- Autoregressive first order (AR (1))

For autoregressive first order (AR (1)), Site and Subject nest within site will be included as random effects (G-side). For the remaining covariance structures only site will be included as a random effect (G-side). The Kenward and Roger method (Kenward and Roger, 1997) will be used for the denominator degree of freedom.

Comparisons between the test and control lens at the 2-weeks follow-up will be carried out using two-sided 95% confidence intervals constructed for least-square mean differences (test

minus control). The lower limit of the 95% confidence interval will be compared to -5 and 0 to test for non-inferiority and superiority, respectively. Non-inferiority of the test lens relative to the control will be concluded if a lower limit is above -5. If non-inferiority is established the superiority will be tested. Superiority will be declared if the lower limit of the 95% confidence interval is above 0.

### 14.6. Secondary Analysis

Not Applicable.

### 14.7. Other Exploratory Analyses

# Driving, Indoor and Outdoor Performance

Each driving, indoor and outdoor performance item will be analyzed separately using a generalized linear mixed model for ordinal data with a multinomial distribution and cumulative logit as a link function. The experimental design factors: sequence of lens wear, period, lens type, first order carryover effect will be included in each model as fixed effects. Site will be included as a random effect. An appropriate covariance structure will be used to model the residual errors between measurements within same subject across study periods.

The assumption of proportionality of odds across response categories will be assessed graphically. If this assumption is violated then the distribution of responses will be investigated. If sparse data is observed then the sparse response categories may be collapsed to ensure there is sufficient data for analysis. If the assumption of proportionality of odds is still violated in the collapsed categories then a partial proportional odds model may be considered. If any of the above models fail to converge, then reduced versions may be considered. A Generalized Estimating Equation (GEE) may also be considered as necessary.

Comparison between the test lens and the control lens at the 2-week follow-up will be carried out using two-sided 95% confidence intervals of the odds ratios (Test over Control); where the odds ratio represents the odds of having a higher positive rating/experience for the Test lens compared to the Control lens.

For driving items, non-inferiority of the test lens relative to the control will be concluded if the lower limit of the 95% confidence interval of the odds ratio is above 0.67. If non-inferiority is met, then superiority will be tested. Superiority of the test lens relative to the control lens will be concluded if the lower limit of the confidence interval of the odds ratio is above 1.

### **CLUE Handling**

CLUE handling will be analyzed and tested in the same exact manner as CLUE comfort and vision as describe above in Section 14.5.

Physiological Responses will be descriptively summarized for each lens type.

### 14.8. Interim Analysis

There will not be an interim analysis performed on this study.

### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 10 imputations.

### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

No external data will be collected of the study.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

# 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the

risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)

- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>15</sup>/Data Protection Act in the United Kingdom<sup>16</sup> /insert applicable country specific regulations and add the appropriate reference in Section 22 and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Ouery resolution
- Case Report Form signature
- Completion of any follow-up action items.

### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

### 22. REFERENCES

- ISO 14155:2011: Clinical investigation of medical devices for human subjects Good clinical practice.
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP).
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. <a href="http://www.wma.net/en/30publications/10policies/b3/index.html">http://www.wma.net/en/30publications/10policies/b3/index.html</a>.
- 4. United States (US) Code of Federal Regulations (CFR).



- 14. Stroup W. Generalized Mixed Models: Modern Concepts, Methods and Applications. 2013 Boca Raton CRC Press. 467-492.
- 15. Health Information Portability and Accountability Act (HIPAA). .
- 16. Data Protection Act.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)

2
10

### APPENDIX B: PATIENT INSTRUCTION GUIDE

A Patient Instruction Guide (PIG) will be provided separately.

### APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

Not Applicable for Investigational Products.

# APPENDIX D: Limbal and Conjunctival (BULBAR) Redness Expanded Sodium Fluorescein Corneal Staining Lens Fitting Characteristics Subject Reported Ocular Symptoms Problems Front and Back Surface Lens Deposit Grading Procedure Determination of Distance Spherocylindrical Refractions Biomicroscopy Scale Distance and Near Visual Acuity Evaluation Patient Reported Outcomes White Light Lens Surface Wettability

### LIMBAL AND CONJUNCTIVAL (BULBAR) REDNESS















### EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING










### LENS FITTING CHARACTERISTICS














### SUBJECT REPORTED OCULAR SYMPTOMS PROBLEMS



# FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE











## DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS

















# **BIOMICROSCOPY SCALE**











CR-6140 v2.0 CONFIDENTIAL Page 118 of 131



# DISTANCE AND NEAR VISUAL ACUITY EVALUATION





## PATIENT REPORTED OUTCOMES



## WHITE LIGHT LENS SURFACE WETTABILITY





#### APPENDIX F: STARTING CONTACT LENS POWER GUIDELINE

| | | Vertexed | Vertexed | Vertexed | Contact |
|--------|----------|----------|----------|----------|---------|
| Sphere | Cylinder | Sphere | Cylinder | SEquiv | Rx |
| -0.75 | -0.50 | -0.743 | -0.497 | -0.992 | -1.00 |
| -0.75 | -0.75 | -0.743 | -0.743 | -1.115 | -1.00 |
| -0.75 | -1.00 | -0.743 | -0.988 | -1.237 | -1.25 |
| -1.00 | 0.00 | -0.988 | 0.000 | -0.988 | -1.00 |
| -1.00 | -0.25 | -0.988 | -0.249 | -1.113 | -1.00 |
| -1.00 | -0.50 | -0.988 | -0.497 | -1.237 | -1.25 |
| -1.00 | -0.75 | -0.988 | -0.743 | -1.360 | -1.25 |
| -1.00 | -1.00 | -0.988 | -0.988 | -1.482 | -1.50 |
| -1.25 | 0.00 | -1.232 | 0.000 | -1.232 | -1.25 |
| -1.25 | -0.25 | -1.232 | -0.249 | -1.356 | -1.25 |
| -1.25 | -0.23 | -1.232 | -0.249 | -1.480 | -1.50 |
| -1.25 | -0.75 | -1.232 | -0.743 | -1.603 | -1.50 |
| -1.25 | | -1.232 | | | -1.75 |
| | -1.00 | | -0.988 | -1.726 | |
| -1.50 | 0.00 | -1.473 | 0.000 | -1.473 | -1.50 |
| -1.50 | -0.25 | -1.473 | -0.249 | -1.598 | -1.50 |
| -1.50 | -0.50 | -1.473 | -0.497 | -1.722 | -1.75 |
| -1.50 | -0.75 | -1.473 | -0.743 | -1.845 | -1.75 |
| -1.50 | -1.00 | -1.473 | -0.988 | -1.968 | -2.00 |
| -1.75 | 0.00 | -1.714 | 0.000 | -1.714 | -1.75 |
| -1.75 | -0.25 | -1.714 | -0.249 | -1.839 | -1.75 |
| -1.75 | -0.50 | -1.714 | -0.497 | -1.963 | -2.00 |
| -1.75 | -0.75 | -1.714 | -0.743 | -2.086 | -2.00 |
| -1.75 | -1.00 | -1.714 | -0.988 | -2.208 | -2.25 |
| -2.00 | 0.00 | -1.953 | 0.000 | -1.953 | -2.00 |
| -2.00 | -0.25 | -1.953 | -0.249 | -2.078 | -2.00 |
| -2.00 | -0.50 | -1.953 | -0.497 | -2.202 | -2.25 |
| -2.00 | -0.75 | -1.953 | -0.743 | -2.325 | -2.25 |
| -2.00 | -1.00 | -1.953 | -0.988 | -2.447 | -2.50 |
| -2.25 | 0.00 | -2.191 | 0.000 | -2.191 | -2.25 |
| -2.25 | -0.25 | -2.191 | -0.249 | -2.315 | -2.25 |
| -2.25 | -0.50 | -2.191 | -0.497 | -2.439 | -2.50 |
| -2.25 | -0.75 | -2.191 | -0.743 | -2.563 | -2.50 |
| -2.25 | -1.00 | -2.191 | -0.988 | -2.685 | -2.75 |
| -2.50 | 0.00 | -2.427 | 0.000 | -2.427 | -2.50 |
| -2.50 | -0.25 | -2.427 | -0.249 | -2.552 | -2.50 |
| -2.50 | -0.50 | -2.427 | -0.497 | -2.676 | -2.75 |
| -2.50 | -0.75 | -2.427 | -0.743 | -2.799 | -2.75 |
| -2.50 | -1.00 | -2.427 | -0.988 | -2.921 | -3.00 |
| -2.75 | 0.00 | -2.662 | 0.000 | -2.662 | -2.75 |
| -2.75 | -0.25 | -2.662 | -0.249 | -2.787 | -2.75 |
| -2.75 | -0.50 | -2.662 | -0.497 | -2.911 | -3.00 |
| -2.75 | -0.75 | -2.662 | -0.743 | -3.034 | -3.00 |
| -2.75 | -1.00 | -2.662 | -0.743 | -3.156 | -3.25 |
| -3.00 | 0.00 | -2.896 | 0.000 | -2.896 | -3.23 |
| -3.00 | -0.25 | -2.896 | -0.249 | -3.020 | -3.00 |
| -3.00 | -0.23 | -2.896 | -0.497 | -3.144 | -3.25 |
| -3.00 | -0.30 | -2.896 | -0.743 | -3.144 | -3.25 |
| -3.00 | -0.75 | -2.896 | -0.743 | -3.390 | -3.50 |
| -3.25 | 0.00 | -3.128 | 0.000 | -3.128 | -3.25 |
| -3.25 | -0.25 | -3.128 | -0.249 | -3.253 | -3.25 |
| -3.25 | -0.50 | -3.128 | -0.497 | -3.377 | -3.50 |
| -3.25 | -0.75 | -3.128 | -0.743 | -3.500 | -3.50 |
| -3.25 | -1.00 | -3.128 | -0.988 | -3.622 | -3.50 |
| -3.50 | 0.00 | -3.359 | 0.000 | -3.359 | -3.25 |
| -3.50 | -0.25 | -3.359 | -0.249 | -3.484 | -3.50 |
| -3.50 | -0.50 | -3.359 | -0.497 | -3.607 | -3.50 |
| -3.50 | -0.75 | -3.359 | -0.743 | -3.731 | -3.75 |

| | | Vertexed | Vertexed | Vertexed | Contact |
|---|---|---|---|---|---|
| Sphere | Cylinder | Sphere | Cylinder | SEquiv | Rx |
| -3.50 | -1.00 | -3.359 | -0.988 | -3.853 | -3.75 |
| -3.75 | 0.00 | -3.589 | 0.000 | -3.589 | -3.50 |
| -3.75 | -0.25 | -3.589 | -0.249 | -3.713 | -3.75 |
| -3.75 | -0.50 | -3.589 | -0.497 | -3.837 | -3.75 |
| -3.75 | -0.75 | -3.589 | -0.743 | -3.960 | -4.00 |
| -3.75 | -1.00 | -3.589 | -0.988 | -4.083 | -4.00 |
| -4.00 | 0.00 | -3.817 | 0.000 | -3.817 | -3.75 |
| -4.00 | -0.25 | -3.817 | -0.249 | -3.941 | -4.00 |
| -4.00 | -0.50 | -3.817 | -0.497 | -4.065 | -4.00 |
| -4.00 | -0.75 | -3.817 | -0.743 | -4.188 | -4.25 |
| -4.00 | -1.00 | -3.817 | -0.988 | -4.311 | -4.25 |
| -4.25 | 0.00 | -4.044 | 0.000 | -4.044 | -4.00 |
| -4.25 | -0.25 | -4.044 | -0.249 | -4.168 | -4.25 |
| -4.25 | -0.50 | -4.044 | -0.497 | -4.292 | -4.25 |
| -4.25 | -0.75 | -4.044 | -0.743 | -4.415 | -4.50 |
| -4.25 | -1.00 | -4.044 | -0.988 | -4.538 | -4.50 |
| -4.50 | 0.00 | -4.269 | 0.000 | -4.269 | -4.25 |
| -4.50 | -0.25 | -4.269 | -0.249 | -4.394 | -4.50 |
| -4.50 | -0.50 | -4.269 | -0.497 | -4.518 | -4.50 |
| -4.50 | -0.75 | -4.269 | -0.743 | -4.641 | -4.75 |
| -4.50 | -1.00 | -4.269 | -0.988 | -4.764 | -4.75 |
| -4.75 | 0.00 | -4.494 | 0.000 | -4.494 | -4.50 |
| -4.75 | -0.25 | -4.494 | -0.249 | -4.618 | -4.50 |
| -4.75 | -0.50 | -4.494 | -0.497 | -4.742 | -4.75 |
| -4.75 | -0.75 | -4.494 | -0.743 | -4.866 | -4.75 |
| -4.75 | -1.00 | -4.494 | -0.988 | -4.988 | -5.00 |
| -5.00 | 0.00 | -4.717 | 0.000 | -4.717 | -4.75 |
| -5.00 | -0.25 | -4.717 | -0.249 | -4.842 | -4.75 |
| -5.00 | -0.50 | -4.717 | -0.497 | -4.965 | -5.00 |
| -5.00<br>-5.00 | -0.75<br>-1.00 | -4.717<br>-4.717 | -0.743<br>-0.988 | -5.089<br>-5.211 | -5.00<br>-5.25 |
| -5.25 | 0.00 | -4.717 | 0.000 | -4.939 | -5.25 |
| -5.25 | -0.25 | -4.939 | -0.249 | -5.063 | -5.00 |
| -5.25 | -0.50 | -4.939 | -0.249 | -5.187 | -5.25 |
| -5.25 | -0.75 | -4.939 | -0.743 | -5.311 | -5.25 |
| -5.25 | -1.00 | -4.939 | -0.988 | -5.433 | -5.50 |
| -5.50 | 0.00 | -5.159 | 0.000 | -5.159 | -5.25 |
| -5.50 | -0.25 | -5.159 | -0.249 | -5.284 | -5.25 |
| -5.50 | -0.50 | -5.159 | -0.497 | -5.408 | -5.50 |
| -5.50 | -0.75 | -5.159 | -0.743 | -5.531 | -5.50 |
| -5.50 | -1.00 | -5.159 | -0.988 | -5.654 | -5.75 |
| -5.75 | 0.00 | -5.379 | 0.000 | -5.379 | -5.50 |
| -5.75 | -0.25 | -5.379 | -0.249 | -5.503 | -5.50 |
| -5.75 | -0.50 | -5.379 | -0.497 | -5.627 | -5.75 |
| -5.75 | -0.75 | -5.379 | -0.743 | -5.751 | -5.75 |
| -5.75 | -1.00 | -5.379 | -0.988 | -5.873 | -5.75 |
| -6.00 | 0.00 | -5.597 | 0.000 | -5.597 | -5.50 |
| -6.00 | -0.25 | -5.597 | -0.249 | -5.722 | -5.75 |
| -6.00 | -0.50 | -5.597 | -0.497 | -5.846 | -5.75 |
| -6.00 | -0.75 | -5.597 | -0.743 | -5.969 | -6.00 |
| -6.00 | -1.00 | -5.597 | -0.988 | -6.091 | -6.00 |
| -6.25 | 0.00 | -5.814 | 0.000 | -5.814 | -5.75 |
| -6.25 | -0.25 | -5.814 | -0.249 | -5.939 | -6.00 |
| -6.25 | -0.50 | -5.814 | -0.497 | -6.062 | -6.00 |
| -6.25 | -0.75 | -5.814 | -0.743 | -6.186 | -6.25 |
| -6.25 | -1.00 | -5.814 | -0.988 | -6.308 | -6.25 |
| -6.50 | 0.00 | -6.030 | 0.000 | -6.030 | -6.00 |

#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6140 / <u>Contact Lenses with New UV-blocker Manufactured with Different Techniques</u>

Version: 2.0, amendment 1 Date: 07 February 2018

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| S | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |